CLINICAL TRIAL: NCT01384240
Title: Evaluation of Low-Cost High Resolution Microendoscope for the Detection of Lower Gastrointestinal Neoplasia
Brief Title: Evaluation of a Low-Cost High Resolution Microendoscope for the Detection of Lower Gastrointestinal Neoplasia
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study is closed as the PI transferred to another institution.
Sponsor: Anandasabapathy, Sharmila, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GCO# 09-1040
Record Dates: First submitted 2011-06-27; First posted 2011-06-29 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Colon Polyps; Colonic Dysplasia; Anal Dysplasia
Keywords: colon polyps; colonic dysplasia; anal dysplasia; microendoscopy
MeSH Terms: conditions — Colonic Polyps | interventions — Proflavine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proflavine Hemisulfate (Experimental)
  Interventions: Drug: Proflavine Hemisulfate

INTERVENTIONS:
Drug: Proflavine Hemisulfate — 3-ml of 0.01% proflavine(derived from dissolving 10 mg proflavine hemisulfate USP in 100 ml sterile water)
  Other Names: Proflavine

SUMMARY:
The overall objective of this study is to obtain data to evaluate whether high-resolution imaging of the colon can assist clinicians in detecting dysplastic (precancerous) and neoplastic areas. This is a pilot study of a novel technology, a miniaturized microscope device which can be used during standard endoscopy to image the gastrointestinal epithelium. Theoretically, by visualizing superficial mucosal changes at a high-resolution and magnification, the investigators will be able to obtain optical images that can be used to guide endoscopic biopsy and polypectomy. This may foster the selective targeting of dysplasia/neoplasia, thereby improving diagnostic accuracy.

ELIGIBILITY:
Inclusion Criteria:

* surveillance of polyps or disease of the colon
* screening colonoscopy
* anoscopy for suspected or known anal dysplasia or neoplasia

Exclusion Criteria:

* unfit for standard colonoscopy or anoscopy
* unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2010-04; Primary Completion 2013-07 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
to determine whether tissue in nepoplastic or non-neoplastic | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Sharmila Anandasabapathy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Chang SS, Shukla R, Polydorides AD, Vila PM, Lee M, Han H, Kedia P, Lewis J, Gonzalez S, Kim MK, Harpaz N, Godbold J, Richards-Kortum R, Anandasabapathy S. High resolution microendoscopy for classification of colorectal polyps. Endoscopy. 2013 Jul;45(7):553-9. doi: 10.1055/s-0032-1326502. Epub 2013 Jun 18. PMID 23780842